CLINICAL TRIAL: NCT00727207
Title: Phase II Trial on Efficacy of mTOR Inhibitor RAD001 as Maintenance Therapy for Patients Above 60 Years in Mantle Cell Lymphoma After First and Second Line Chemotherapy
Brief Title: Everolimus in Treating Older Patients With Mantle Cell Lymphoma Previously Treated With First-Line or Second-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of participations (8 of 25)
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000597004; KRDI-TUM-CRAD001C2428; EUDRACT: 2007-005116-12; EU-20855
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well everolimus works in treating older patients with mantle cell lymphoma who received previous first-line or second-line chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of older patients with mantle cell lymphoma receiving everolimus and who were previously treated with first- or second-line chemotherapy.

Secondary

* Determine the toxicity and feasibility of treatment with this drug.
* Determine the efficacy of this drug in these patients.
* Compare the duration of remission after first- vs second-line chemotherapy.
* Determine the rate of objective remission.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of mantle cell lymphoma
* Stable disease after first- or second-line chemotherapy
* No uncontrolled cerebral or leptomeningeal disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* Age ≥ 60 years or patients ≥ 40 and < 60 years who are not suitable for high-dose chemotherapy followed by autologous stem cell transplantation or allogeneic stem cell transplantation
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* SGPT and SGOT ≤ 3 times ULN
* Bilirubin ≤ 1.5 times ULN
* No other malignancies within the past 3 years except treated cervical carcinoma or basal cell cancer
* No other serious or non-controlled illnesses (e.g., diabetes mellitus, uncontrolled hypertension, serious infections, serious malnutrition, unstable angina pectoris, weak heart, myocardial infarction within the past 6 months, chronic liver illness, active ulceration in the gastrointestinal tract, psychiatric illness)
* No known HIV infection
* No gastrointestinal disturbances that could influence the absorption of everolimus and cause short-intestine syndrome (e.g., atrophic gastritis)
* No coagulation or bleeding diatheses
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Patients must have complied with their previous drug prescription

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* See Patient Characteristics
* Recovered from all prior therapy
* At least 2 weeks since prior surgery, radiotherapy, or systemic antitumor therapy
* More than 4 weeks since prior experimental medication
* No chronic therapy with systemic steroids or other immunosuppressants except rituximab
* No prior organ transplantation
* No therapy with vitamin K antagonist, except low-dose coumarin
* No prior mTOR inhibitors

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Toxicity and feasibility
Efficacy
Comparison of duration of remission after first- vs second-line chemotherapy
Rate of objective remission

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keller, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich, Germany